CLINICAL TRIAL: NCT04639349
Title: Effect of Home Exercise Activity on Cortisol and Depression in COPD Patients During the Pandemic COVID-19
Brief Title: Effect of Home Exercise Activity on Cortisol and Depression in COPD During the Pandemic COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002897
Record Dates: First submitted 2020-11-19; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercised group (Experimental): the exercise group (20 patients) will receive a exercise session contains a fifty minutes exercise training at home with moderate intensity on the available training devices as bicycle or treadmill in addition to 30 minutes of exercising of upper and lower limb, the session will be repeated three times per week for eight weeks.
  Interventions: Behavioral: exercise group
- control group (Other): The control group will not be trained
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: exercise group — the exercise group (20 patients) will receive a exercise session contains a fifty minutes exercise training at home with moderate intensity on the available training devices as bicycle or treadmill in addition to 30 minutes of exercising of upper and lower limb, the session will be repeated three times per week for eight weeks.
  Arms: Exercised group
Other: control group — the control group will not be trained
  Arms: control group

SUMMARY:
exercise activity during the COVID pandemic is appreciated to be conducted in home especially for chronic chest diseases as chronic obstructive pulmonary disease (COPD) to reduce the chance of viral contamination during the COVID-19 pandemic.

DETAILED DESCRIPTION:
40 COPD men will be divided to exercise group (20 patients) and control group (20 patients):

the exercise group will receive a exercise session contains a fifty minutes exercise training at home with moderate intensity on the available training devices as bicycle or treadmill in addition to 30 minutes of exercising of upper and lower limb, the session will be repeated three times per week for eight weeks.

The control group will not be trained

ELIGIBILITY:
Inclusion Criteria:

* stable COPD patients
* patients who will have a training device as bicycle or treadmill in home

Exclusion Criteria:

* diabetic patients
* renal patients.
* liver diseases

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 40 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
cortisol | It will be measured after eight weeks of training
  it will be measured in plasma
hospital anxiety and depression scale | It will be measured after eight weeks of training
  this a questionnaire that will assess anxiety and depression in COPD patients

SECONDARY OUTCOMES:
pulmonary function test | It will be measured after eight weeks of training
  it will be a measurement for lung volume and capacities
Interleukin-8 | It will be measured after eight weeks of training
  It is an inflammatory marker in plasma
body mass index | It will be measured after eight weeks of training
  it will measure body mass changes
six minute walking test | It will be measured after eight weeks of training
  it assess functional capacity
St. George's respiratory questionnaire | It will be measured after eight weeks of training
  It assess the effect of COPD on general quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt